CLINICAL TRIAL: NCT02954055
Title: A Randomized Phase II Trial of Metronomic Oral Vinorelbine Plus Cyclophosphamide and Capecitabine (VEX) Versus Weekly Paclitaxel as First-line or Second-line Treatment in Patients With ER-positive/HER2-negative Advanced or Metastatic Breast Cancer
Brief Title: MEtronomic TrEatment Option in Advanced bReast cAncer
Acronym: METEORA-II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCSG 54-16; 2016-002200-39 (EudraCT Number)
Record Dates: First submitted 2016-09-26; First posted 2016-11-03 (Estimated); Results first posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: locally advanced; metastatic; breast cancer; ER-positive; HER2-negative; Stage IV
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Paclitaxel; Cyclophosphamide; Capecitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Paclitaxel 90 mg/m2 days 1, 8, 15 q4w. Patients will continue to receive assigned treatment until progression or lack of tolerability.
  Interventions: Drug: Paclitaxel
- Arm B (Experimental): Metronomic VEX:
  Cyclophosphamide 50 mg orally once daily continuously, Capecitabine 500 mg, orally 3 times a day (1500 mg/day) continuously, Vinorelbine 40 mg orally days 1, 3, 5 each week continuously. Patients will continue to receive assigned treatment until progression or lack of tolerability.
  Interventions: Drug: Cyclophosphamide; Drug: Capecitabine; Drug: Vinorelbine

INTERVENTIONS:
Drug: Paclitaxel — Arm A
  Other Names: Paclitaxel Sandoz
  Arms: Arm A
Drug: Cyclophosphamide — Arm B
  Other Names: Endoxan Baxter
  Arms: Arm B
Drug: Capecitabine — Arm B
  Other Names: Xeloda
  Arms: Arm B
Drug: Vinorelbine — Arm B
  Other Names: Navelbine
  Arms: Arm B

SUMMARY:
This is a multi-center, randomized phase II trial that will randomise women with ER-positive, HER2-negative (Human Epidermal Growth factor Receptor 2-negative) metastatic or locally relapsed breast cancer in a ratio of 1:1 to receive a metronomic regimen of vinorelbine plus cyclophosphamide and capecitabine, or the conventional paclitaxel monotherapy.

DETAILED DESCRIPTION:
The prognosis for patients with locally advanced or metastatic disease (ABC) remains poor, with a median survival of 2-4 years. About 10% of newly diagnosed BC patients present with ABC, and 30% to 50% of patients diagnosed at earlier stages will subsequently develop metastatic disease.

In the first-line treatment of HER2 (Human Epidermal Growth factor Receptor 2) negative ABC patients, various chemotherapy regimens can be used including taxanes, which are among the most active agents in BC. Single agent response rates range from 20 to 50%. However, eventually all patients will progress with a median time to progression of 5 to 7 months. A weekly (qw) over a three-weekly (q3w) administration schedule of paclitaxel has been shown to be more effective in the metastatic as well as in the adjuvant setting after standard chemotherapy

The VEX regimen was recently investigated within a phase II trial currently ongoing at the European Institute of Oncology (IEO) (IEO number IEOS582/111; EudraCT Number: 2010-024266-21; title: "A phase II study of metronomic oral chemotherapy with cyclophosphamide plus capecitabine and vinorelbine in metastatic breast cancer patients"). Patients received vinorelbine 40 mg orally on days 1, 3 and 5 every week, cyclophosphamide 50 mg daily and capecitabine 500 mg 3 times a day.

Given the promising activity of the VEX regimen in a pre-treated population of advanced breast cancer patients and the good tolerability, the aim of the present trial is to investigate whether the VEX schedule may improve efficacy and tolerability as compared to standard paclitaxel treatment in advanced or metastatic ER-positive/HER2-negative breast cancer patients.

The concept of the VEX metronomic treatment is to administer the combination for as long as the patient has the possibility of deriving a benefit from it. The time to treatment failure (TTF) has been chosen as primary endpoint for this trial. TTF is defined as time from the date of randomization to the date when the final dose of trial treatment is administered. Chemotherapy may need to be stopped due to lack of tolerability, lack of efficacy or patient preference through subjective symptom assessment. TTF is a composite endpoint combining all these feasibility aspects of a treatment. It is therefore uniquely suited to the research question of the current trial. The secondary endpoints progression-free survival, disease control and safety will allow further assessment of the feasibility of the VEX metronomic treatment versus the paclitaxel monotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed HER2-negative locally advanced or metastatic (stage IV) breast cancer.
* Maximum of one prior line of chemotherapy for advanced or metastatic breast cancer.
* Measurable or non-measurable, but radiologically evaluable (except for skin lesions), disease according to RECIST 1.1 criteria.
* Female aged 18 years or older.
* Life expectancy > 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* ER-positive disease by local laboratory, determined on most recent available tissue (latest biopsy of metastatic lesion, otherwise prior biopsy or surgical specimen).
* If previously treated with a taxane in the neoadjuvant or adjuvant setting, the period from end of treatment to disease recurrence must have been > 12 months (> 365 days).
* Radiation therapy, if given and regardless of site, must be completed at least 2 weeks prior to randomization.
* Normal hematologic status,
* Absolute neutrophil count ≥1000/mm3 (1.0 × 109/L),
* Platelets ≥ 100 × 109/L,
* Hemoglobin ≥ 9 g/dL (≥ 90 g/L).
* Normal renal function: serum creatinine ≤ 1.5 ULN or calculated creatinine clearance ≥ 50 mL/min according to the Cockcroft-Gault formula.
* Normal liver function:
* Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN). In the case of known Gilbert's syndrome, a higher serum total bilirubin (< 3 × ULN) is allowed.
* Aspartate transaminase (AST) and Alanine transaminase (ALT) ≤ 3 × ULN; if the patient has liver metastases, ALT and AST must be ≤ 5 × ULN.
* Women of child bearing potential must have documented negative pregnancy test within 2 weeks prior to randomization and agree to acceptable birth control (non-hormonal) during and up to 6 months after trial therapy.
* Written Informed Consent (IC) must be signed and dated by the patient and the Investigator prior to starting screening procedures and randomization.
* The patient has been informed of and agrees to data transfer and handling, in accordance with national data protection guidelines.

Exclusion Criteria:

* More than one prior line of chemotherapy for advanced or metastatic breast cancer
* Previous treatment for advanced or metastatic disease with taxanes, or capecitabine or vinorelbine or oral cyclophosphamide.
* More than 2 lines of previous endocrine therapy for locally advanced or metastatic breast cancer.
* Known active central nervous system metastases, as indicated by clinical symptoms, cerebral edema, and/or progressive growth (patients with history of Central Nervous System (CNS) metastases or spinal cord compression are eligible if they are clinically and radiologically stable for at least 4 weeks before first dose of trial treatment and have not required high-dose steroid treatment in the last 4 weeks).
* Peripheral neuropathy grade 2 or higher (CTCAE version 4.0).
* Significant uncontrolled cardiac disease (i.e. unstable angina, myocardial infarction within prior 6 months), patients classified as having a New York Heart Association (NYHA) class III or IV congestive heart failure.
* Pregnant or lactating.
* Prior history of non-breast malignancy (except for adequately controlled basal cell carcinoma of the skin, carcinoma in situ of the cervix, in situ carcinoma of the bladder).
* Any concurrent condition which in the Investigator's opinion makes it inappropriate for the patient to participate in the trial or which would jeopardize compliance with the protocol.
* Contraindications or known hypersensitivity to the trial medication or excipients.
* The use of any anti-cancer investigational agents within 30 days prior to expected start of trial treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2022-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Munzone, MD, Study Chair — European Institute of Oncology
Locations (20):
- Italy (20):
  - Centro di Riferimento Oncologico (CRO), Aviano
  - A.O.U. di Bologna Policlinico S. Orsola-Malpighi Viale Ercolani 4/2, Bologna
  - Ospedale di Bolzano Oncologia Medica Via lorenz Bohler 5, Bolzano
  - Aziendale Spedali Civili di Brescia SSVD Breast Unit P.le Spedali Civili 1, Brescia
  - "Antonio Perrino" Division of Medical Oncology Strada Statale 7 APPIA, Brindisi
  - Candiolo Cancer Institute (FPO-IRCCS), Candiolo
  - ASST Di Cremona, Unità di Patologia Mammaria-Breast Unit VIALE CONCORDIA 1, Cremona
  - Ospedale Misericordia di Grosseto, Grosseto
  - ASST Ovest Milanese Oncology Department Via Papa Giovanni Paolo II, Legnano
  - Ospedale Generale Provinciale di Macerata, Macerata
  - IRST IRCCS Division of medical oncology Via Maroncelli 40, Meldola
  - Istituto Europeo di Oncologia, Division of Medical Senology, Via Ripamonti 435, Milan
  - Osp. Sacro Cuore Don Calabria Division in Medical Oncology, Negrar
  - Istituti Clinici Scientifici Maugeri SpA SB, Pavia
  - Ospedale S. Maria delle Croci, Ravenna
  - Ospedale Infermi Uo Oncologia Via Settembrini 2, Rimini
  - Fondazione Policlinico Universitario A.Gemelli, Rome
  - A.O.U Città della Salute e della Scienza di Torino SSCVD Oncologia Medica Senologica (Oncology Dep.- Breast Unit) Via Cherasco 23, Torino
  - Asst Bg Ovest Ospedale Di Treviglio, Treviglio
  - ASST Settelaghi - Ospedale di Circolo e Fondazione Macchi U.O Oncologia Medica Viale L. Borri, 57, Varese

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sotiriou C, Pusztai L. Gene-expression signatures in breast cancer. N Engl J Med. 2009 Feb 19;360(8):790-800. doi: 10.1056/NEJMra0801289. No abstract available. PMID 19228622
- [Background] Senkus E, Cardoso F, Pagani O. Time for more optimism in metastatic breast cancer? Cancer Treat Rev. 2014 Mar;40(2):220-8. doi: 10.1016/j.ctrv.2013.09.015. Epub 2013 Oct 1. PMID 24126121
- [Background] Eniu A, Palmieri FM, Perez EA. Weekly administration of docetaxel and paclitaxel in metastatic or advanced breast cancer. Oncologist. 2005 Oct;10(9):665-85. doi: 10.1634/theoncologist.10-9-665. PMID 16249346
- [Background] Miller K, Wang M, Gralow J, Dickler M, Cobleigh M, Perez EA, Shenkier T, Cella D, Davidson NE. Paclitaxel plus bevacizumab versus paclitaxel alone for metastatic breast cancer. N Engl J Med. 2007 Dec 27;357(26):2666-76. doi: 10.1056/NEJMoa072113. PMID 18160686
- [Background] Miles DW, Chan A, Dirix LY, Cortes J, Pivot X, Tomczak P, Delozier T, Sohn JH, Provencher L, Puglisi F, Harbeck N, Steger GG, Schneeweiss A, Wardley AM, Chlistalla A, Romieu G. Phase III study of bevacizumab plus docetaxel compared with placebo plus docetaxel for the first-line treatment of human epidermal growth factor receptor 2-negative metastatic breast cancer. J Clin Oncol. 2010 Jul 10;28(20):3239-47. doi: 10.1200/JCO.2008.21.6457. Epub 2010 May 24. PMID 20498403
- [Background] Seidman AD, Berry D, Cirrincione C, Harris L, Muss H, Marcom PK, Gipson G, Burstein H, Lake D, Shapiro CL, Ungaro P, Norton L, Winer E, Hudis C. Randomized phase III trial of weekly compared with every-3-weeks paclitaxel for metastatic breast cancer, with trastuzumab for all HER-2 overexpressors and random assignment to trastuzumab or not in HER-2 nonoverexpressors: final results of Cancer and Leukemia Group B protocol 9840. J Clin Oncol. 2008 Apr 1;26(10):1642-9. doi: 10.1200/JCO.2007.11.6699. PMID 18375893
- [Background] Sparano JA, Wang M, Martino S, Jones V, Perez EA, Saphner T, Wolff AC, Sledge GW Jr, Wood WC, Davidson NE. Weekly paclitaxel in the adjuvant treatment of breast cancer. N Engl J Med. 2008 Apr 17;358(16):1663-71. doi: 10.1056/NEJMoa0707056. PMID 18420499
- [Derived] Munzone E, Regan MM, Cinieri S, Montagna E, Orlando L, Shi R, Campadelli E, Gianni L, Palleschi M, Petrelli F, Bengala C, Generali D, Collova E, Puglisi F, Cretella E, Zamagni C, Chini C, Ruepp B, Loi S, Colleoni M; International Breast Cancer Study Group (IBCSG). Efficacy of Metronomic Oral Vinorelbine, Cyclophosphamide, and Capecitabine vs Weekly Intravenous Paclitaxel in Patients With Estrogen Receptor-Positive, ERBB2-Negative Metastatic Breast Cancer: Final Results From the Phase 2 METEORA-II Randomized Clinical Trial. JAMA Oncol. 2023 Sep 1;9(9):1267-1272. doi: 10.1001/jamaoncol.2023.2150. PMID 37440239

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Paclitaxel 90 mg/m2 days 1, 8, 15 q4weeks. Patients will continue to receive assigned treatment until progression or lack of tolerability.
  Paclitaxel: Arm A
- Arm B: Metronomic VEX:
  Cyclophosphamide 50 mg orally once daily continuously, capecitabine 500 mg, orally 3 times a day (1500 mg/day) continuously, vinorelbine 40 mg orally days 1, 3, 5 each week continuously. Patients will continue to receive assigned treatment until progression or lack of tolerability.
  Cyclophosphamide: Arm B
  Capecitabine: Arm B
  Vinorelbine: Arm B
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 69 | 71
Completed | 63 | 70
Not Completed | 6 | 1
Not completed — Did not initiate therapy | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Paclitaxel 90 mg/m2 days 1, 8, 15 q4weeks. Patients continued to receive assigned treatment until objective progressive disease (PD), symptomatic deterioration, unacceptable toxicity, death, or refusal to continue treatment, whichever occurred first.
  Paclitaxel: Arm A
- Arm B: Metronomic VEX:
  Cyclophosphamide 50 mg orally once daily continuously, capecitabine 500 mg, orally 3 times a day (1500 mg/day) continuously, vinorelbine 40 mg orally days 1, 3, 5 each week continuously. Patients continued to receive assigned treatment until objective progressive disease (PD), symptomatic deterioration, unacceptable toxicity, death, or refusal to continue treatment, whichever occurred first.
  Cyclophosphamide: Arm B
  Capecitabine: Arm B
  Vinorelbine: Arm B
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 63 | 70 | 133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 47 | 88
  >=65 years | 22 | 23 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 70 | 133
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 63 | 70 | 133

OUTCOME MEASURES:

1. Primary Outcome: Time to Treatment Failure (TTF) Compared Between Treatment Groups.
Description: Efficacy and tolerability, measured by time to treatment failure, of metronomic oral vinorelbine plus cyclophosphamide and capecitabine (VEX) versus weekly paclitaxel, using an intent-to-treat analysis approach.
Time Frame: Assessed at the start of every 4-week (28-day) treatment cycle from randomization to the end of treatment date or discontinuation; median follow-up was 29 months, with a minimum of 0.2 months and maximum of 48.5 months.
Measure: Median (Standard Error); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 63 | 70
months | 5.7 (0.06) | 8.3 (0.06)

2. Secondary Outcome: Frequency of Targeted Adverse Events (Safety and Tolerability).
Description: Frequency of adverse events by type and worst grade experienced.
Time Frame: Time from day 1 of cycle 1 until 28 days after stopping trial treatment.
Reporting Status: Not Posted

3. Secondary Outcome: Disease Control
Description: Defined as best overall response of complete response (CR) or partial response (PR), or stable disease (SD) (or non-CR/non-PD in the case of non-measurable disease only) lasting for at least 24 weeks (at least 2 scans), measured from randomization until first documentation of progressive disease. Best overall response was defined as best response recorded from randomization across all time points until disease progression. Confirmation of partial or complete response by an additional scan was not requested in this trial. Disease response and progression were assessed according to the revised Response Evaluation Criteria in Solid Tumors (RECIST version 1.1)
Time Frame: Tumor measurements were assessed at baseline, and every 12 weeks (± 2 weeks) from randomization until first disease progression on the basis of clinical and radiological tumor assessments, on average approximately 9 months.
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 63 | 70
participants
  Complete response (CR) | 1 | 1
  Partial response (PR) | 18 | 22
  Stable disease (SD)/non-complete response (CR)/non-progressive disease (PD) | 25 | 32
  Progressive disease (PD) | 18 | 11
  Not evaluable (NE) | 1 | 4

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from randomization until documented disease progression according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria or death, whichever occurred first; the death must have occurred within an interval of time corresponding to the interval of tumor re-evaluations. For patients without progression, follow-up was censored at the date of last disease assessment.
Time Frame: as for outcome 3
Measure: Median (Standard Error); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 63 | 70
months | 6.9 (0.06) | 11.1 (0.05)

5. Secondary Outcome: Overall Survival
Description: Overall survival from time of randomisation will be summarised for each treatment group.
Time Frame: From day 1 of cycle 1 until death from any cause (censored at date of last assessment of vital status for patients lost to follow up), assessed up to 36 months from the enrollment of the first patient.
Measure: Median (Standard Error); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 63 | 70
months | 33.7 (0.03) | 29.5 (0.03)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from the first dose of trial medication, at day 1 of every treatment cycle, until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication. In the absence of tumor progression, the patient continued to be followed for SAE reporting according and for documented disease progression or a maximum of 12 months after treatment stop, up to approximately 49 months.
Description: AEs were collected from the first dose of trial medication until 28 days after all treatment discontinuation (EOT visit), regardless of whether it is considered related to a medication. The main criterion for tolerability is the occurrence of toxicities and adverse events. The severity and causality classified according to the NCI CTCAE Version 4.0.
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 1/63 | 3/70
Serious Adverse Events (participants affected / at risk) | 18/63 | 31/70
Other Adverse Events (participants affected / at risk) | 63/63 | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=63) | Arm B (N=70)
Anemia (Blood and lymphatic system disorders) | 2 | 5 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 4 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Anaphylaxis (Immune system disorders) | 1 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Allergic reaction (Immune system disorders) | 1 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Anorexia (Metabolism and nutrition disorders) | 0 | 1 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Diarrhea (Gastrointestinal disorders) | 0 | 1 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Constipation (Gastrointestinal disorders) | 0 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Mucositis oral (Gastrointestinal disorders) | 0 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Nausea (Gastrointestinal disorders) | 0 | 2 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Vomiting (Gastrointestinal disorders) | 0 | 2 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Infection (Infections and infestations) | 0 | 1 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Arthralgia and/or myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Injection site reaction (General disorders) | 0 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Fatigue (General disorders) | 0 | 4 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Acute coronary syndrome (Cardiac disorders) | 0 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Sinus brachycardia (Cardiac disorders) | 0 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Optic nerve disorder (Nervous system disorders) | 0 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Neutrophil count decreased (Blood and lymphatic system disorders) | 8 | 20 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Aspartate aminotransferase increased (Immune system disorders) | 0 | 3 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Pulmonary valve disease (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Alkaline phosphatase increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 12
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=63) | Arm B (N=70)
Anemia (Blood and lymphatic system disorders) | 41 | 26 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Alopecia (Skin and subcutaneous tissue disorders) | 21 | 2 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 5 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Anaphylaxis (Immune system disorders) | 1 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Allergic reaction (Immune system disorders) | 6 | 2 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Anorexia (Metabolism and nutrition disorders) | 1 | 5 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Diarrhea (Gastrointestinal disorders) | 12 | 22 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Constipation (Gastrointestinal disorders) | 13 | 6 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Mucositis oral (Gastrointestinal disorders) | 7 | 5 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
nausea (Gastrointestinal disorders) | 17 | 30 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Vomiting (Gastrointestinal disorders) | 9 | 8 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Peripheral sensory neuropathy (Nervous system disorders) | 30 | 5 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Infection (Infections and infestations) | 20 | 14 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Arthralgia and/or myalgia (Musculoskeletal and connective tissue disorders) | 22 | 20 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Injection site reaction (General disorders) | 2 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Fatigue (General disorders) | 36 | 31 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Acute coronary syndrome (Cardiac disorders) | 1 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Sinus brachycardia (Cardiac disorders) | 0 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Supraventricular tachycardia (Cardiac disorders) | 3 | 4 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Optic nerve disorder (Nervous system disorders) | 1 | 2 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 10 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Neutrophil count decreased (Blood and lymphatic system disorders) | 13 | 11 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Asparate aminotransferase increased (Immune system disorders) | 19 | 14 — Adverse events were collected from the first dose of trial medication until 28 days after all treatment discontinuation (end of treatment visit), regardless of whether it is considered related to a medication.
Aortic valve disease (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 2
Sudden death, not otherwise specified (General disorders) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
GGT increased (Investigations) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Facial nerve disorder (Nervous system disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT02954055/Prot_SAP_000.pdf